CLINICAL TRIAL: NCT01549756
Title: Qualitative Research for Stage 4 Stomach Cancer and Their Caregivers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Find A Cure Panel (Other)
Responsible Party: Sponsor
Other Study IDs: facpsc1001
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Stage 4 Stomach/Gastric Cancer; Patients and Caregivers
Keywords: stage 4 stomach cancer; stage 4 gastric cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Qualitative Research: Experiential/opinion based research
  Interventions: Behavioral: bulletin board and teleophone depth interview

INTERVENTIONS:
Behavioral: bulletin board and teleophone depth interview — qualitative based research

SUMMARY:
Find A Cure Panel is looking for people with Stage 4 stomach/gastric cancer or the caregivers of people with Stage 4 stomach/gastric cancer to participate in anonymous and qualitative research that will take an estimated 60 minutes of your time.

This is opinion based, experiential research and is NOT a drug trial.

Note that Stage IV is also known as "advance disease" or metastatic stomach/gastric cancer.

If you are interested in participating, please email FACP at: info@findacurepanel.com

ELIGIBILITY:
Inclusion Criteria:stage 4 stomach cancer patients and caregivers -

Exclusion Criteria:loved one must still be living

-

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stage 4 stomach cancer patients and caregivers
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-04 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Sample Czar, Los Angeles, California, United States

REFERENCES:
- See also: Related Info — http://www.findacurepanel.com